CLINICAL TRIAL: NCT07197411
Title: A Comparative Study of Portable Patch-type Carotid Ultrasound CADFlow and Desktop Ultrasound Machines
Status: Not yet recruiting | Type: Observational
Sponsor: Xuzhou Medical University Affiliated Suqian Hospital (Other)
Responsible Party: Principal Investigator, Ming, Sun, Xuzhou Medical University Affiliated Suqian Hospital, Xuzhou Medical University Affiliated Suqian Hospital
Other Study IDs: 202509141301
Record Dates: First submitted 2025-09-14; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Device Replacement
MeSH Terms: interventions — Hemodynamic Monitoring

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cohort of healthy adults: Monitoring hemodynamic parameters in healthy subjects using two distinct devices
  Interventions: Diagnostic Test: Evaluating the Consistency and Accuracy of Two Devices in Monitoring Hemodynamic Parameters; Device: Hemodynamic monitoring

INTERVENTIONS:
Diagnostic Test: Evaluating the Consistency and Accuracy of Two Devices in Monitoring Hemodynamic Parameters — This portable patch-type carotid ultrasound has not yet been used in clinical settings.
Device: Hemodynamic monitoring — Whether the parameters monitored by portable patch-based ultrasound devices agree with the gold standard has not yet been thoroughly validated

SUMMARY:
observational study The purpose of this observational study is to clarify the consistency, accuracy, and reproducibility of portable patch carotid ultrasound (CADFlow) compared to desktop ultrasound machines in detecting cardiac output (CO), peak velocity (Vmax), and minimum velocity (Vmin) in healthy volunteers.

DETAILED DESCRIPTION:
Parameters including cardiac output (CO), peak carotid artery velocity (Vmax), and minimum velocity (Vmin) were monitored in healthy subjects using a portable patch-type carotid ultrasound device (CADFlow). The subjects were placed in a supine position with the head rotated 30° to the contralateral side and the neck slightly extended. The dual-patch probe was then attached to the sites of the most prominent bilateral carotid artery pulsations. The automatic measurement mode was initiated to record blood flow waveforms for 60 seconds. After 30 minutes, the same subjects underwent reassessment of the aforementioned parameters using a conventional ultrasound system. The distal internal diameters of the bilateral common carotid arteries were measured in two-dimensional mode (mean of three measurements). Using pulsed-wave Doppler with an insonation angle ≤60°, Vmax and Vmin were recorded over three consecutive cardiac cycles. The probe was subsequently switched to a transthoracic cardiac probe for CO measurement at the left ventricular outflow tract (LVOT) (mean of three consecutive measurements). The order in which the subjects were monitored with the two devices was randomized.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 79 years; No abnormalities found in physical examination; Signed informed consent form.

Exclusion Criteria:

* Previous or current cardiovascular or cerebrovascular diseases; Carotid intima-media thickness (IMT) ≥ 1.0 mm or plaque; Arrhythmia; ④ BMI > 35 kg/m²; Pregnancy.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Include healthy individuals aged 18 to 79
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Consistency Between Two Devices | through study completion, an average of six months
  Hemodynamic parameters, including cardiac output (CO), peak carotid artery velocity (Vmax), and minimum velocity (Vmin), were monitored in healthy subjects using both a portable patch-based ultrasound device and a conventional console ultrasound machine. The agreement and accuracy between the two devices were evaluated by comparing the correlation coefficients of the parameters and analyzing the mean bias using Bland-Altman plots

CONTACTS AND LOCATIONS:
Locations (1):
- Xuzhou Medical University Affiliated Suqian Hospital, Suqian, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No